CLINICAL TRIAL: NCT04371406
Title: Efficacy of Azithromycin-associated Hydroxychloroquine Therapy Given in General Practice in Early-stage Disease in COVID-19 Patients: Randomized Controlled Trial: MG-COVID
Brief Title: Efficacy of Azithromycin-associated Hydroxychloroquine Therapy Given in General Practice in Early-stage Disease in COVID-19 Patients
Acronym: MG-COVID
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Regulatory approvals have not been obtained
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200447; 2020-001702-35 (EudraCT Number)
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: Covid-19; hydroxychloroquine; primary care; azithromycin
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Hydroxychloroquine sulfate (PLAQUENIL®), 200mg x 3 /d, for 10 days AND Azithromycin (ZITHROMAX®), 500mg on D1 and then 250mg/d for the next 4 days, in addition to standard of care
  Interventions: Drug: Hydroxychloroquine and Azithromycin
- Control Arm (Sham Comparator): Dietetary supplement, Azinc form and vitality®, 2 capsules per day, for 10 days, in addition to standard of care
  Interventions: Dietary Supplement: Azinc

INTERVENTIONS:
Drug: Hydroxychloroquine and Azithromycin — Hydroxychloroquine sulfate (PLAQUENIL®), 200mg x 3 /d, for 10 days AND Azithromycin (ZITHROMAX®), 500mg on D1 and then 250mg/d for the next 4 days, in addition to standard of care
  Arms: Experimental Arm
Dietary Supplement: Azinc — Dietetary supplement, Azinc form and vitality®, 2 capsules per day, for 10 days, in addition to standard of care
  Arms: Control Arm

SUMMARY:
Hydroxychloroquine, a derivative of chloroquine (an antimalarial drug) with a weak immunosuppressive effect, is prescribed by some teams alone or in combination with azithromycin. No randomized controlled trials have demonstrated its efficacy, particularly in primary care in the early stages of the disease. However, currently available data suggest better efficacy if treatment is given early in the disease, before symptoms worsen. To date, the majority of COVID-19 patients treated in outpatient care, particularly in general practice, represent the majority of COVID-19 patients.

It is essential to evaluate, in primary care, the efficacy and safety of hydroxychloroquine combined with azithromycin in Covid-19 patients in order to be able to implement this therapeutic strategy as soon as the first symptoms appear. We realize a randomized, controlled, open superiority trial, in 2 parallel groups (ratio 1:1).The main objective is to assess the efficacy of Hydroxychloroquine combined with azithromycin in COVID-19 patients in primary care, in add-on to standard of care, on unfavorable outcome defined by the onset of at least one of the following between D0 and D14: hospitalization, death or percutaneous O² saturation ≤ 92% in ambient air.

DETAILED DESCRIPTION:
Randomized, controlled, open superiority trial, in 2 parallel groups (ratio 1:1).

Eligible consecutive patient will be offered to take part in the trial during a visit to thier GP for COVID symptoms. After verification of eligibility criteria and written informed consent, a nasopharyngeal swab, an ECG and a blood sampled (kalaemia, magnesemia and calcemia) will be performed.

Patient with SARS-CoV-2 PCR positive result and still fulfilling eligibility criteria will be randomized on day2 (D2) through a web-based allocation system, following a computer generated allocation list, stratified on center and existence of any comorbidity, to experimental or control group. Patients without confirmation of SARS-CoV-2 infection on PCR will not continue the trial. Both groups patients will have a paper-based diary to record their daily symptoms and drug intake. A clinical follow-up will be done by the GP at D5, D8, D14 and D28.The main analysis population will be in intention to treat. An intermediate efficacy analysis is planned when 50% of patients have reached D14.

Two hundred consecutive patients (from pre-identified centers) will be included in an ancillary virological study to assess evolution of viral load at D8 and D14. For these patients all nasopharyngeal swab will be sent to a centralised lab at Pitié-Salpêtrière Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria :
* Adult aged 18 to 75 years old
* Taken into primary health care for suspicion of early-stage COVID-19 infection (maximum 5 days of evolution). The patient must have presented within the previous 5 days at least one of the following criteria: fever (≥38°C), cough, anosmia, agueusia, diarrhea, headache, myalgia.

Criteria for randomization at D2 :

* Positive PCR on deep nasopharyngeal swab.
* Kalemia ≥ 3.5 mmol/L
* Normal magnesium and calcium levels (according to laboratory standards)
* QTc ≤ 460ms for women or QTc ≤ 450ms for men
* Beta-hCG negative

Exclusion criteria :

* Comorbidity(ies) or clinical condition of the patient requiring immediate oxygen therapy, hospitalization and/or ventilatory assistance
* Concomitant treatment contraindicated, not recommended, or with precautions for use in combination with hydroxychloroquine or azithromycin:

  * drug likely to induce torsades de pointe or at increased risk of ventricular arrhythmia, and in particular citalopram, escitalopram, hydroxyzine, domperidone, piperazine, class IA and III antiarrhythmics, tricyclic antidepressants, antipsychotics and certain anti-infectives (macrolides, fluoroquinolones).
  * Alkaloids of ergot of rye, colchicine, cisapride
  * proconvulsant or epileptogenic threshold lowering drugs: imipraminic antidepressants, selective serotonin reuptake inhibitors, neuroleptics (phenothiazines and butyrophenones) and tramadol.
* Known history of contraindications or increased risk of treatment with hydroxychloroquine or azithromycin (retinopathy,renal failure, significant liver failure, severe cholestasis, porphyria, known G6PD deficit, hypomagnesemia and hypokalemia, diabetes, myasthenia gravis, Heart diseases (heart failure, infarction, arrhythmia, congenital QTc prolongation, abnormalities that interfere with QTc measurement such as Left Bundle Branch Block, Right Bundle Branch Block, Pace maker with ventricular pacing), epilepsy, allergy to hydroxychloroquine, chloroquine, azithromycin, erythromycin, any other macrolide, ketolide or any of the excipients of Plaquenil® or Zithromax® or any of the components of Azinc form and vitality®.
* Ongoing treatment with hydroxychloroquine or azithromycin, regardless of the indication.
* Taking other antiviral targeted therapy used in COVID-19 disease
* Women who are pregnant or breastfeeding or planning to become pregnant within 8 months of discontinuing hydroxychloroquine therapy.
* No National Health Insurrance (sécurité sociale, CMU or AME) coverage.
* Major under guardianship or curatorship
* Participation in another therapeutic clinical trial for COVID-19
* Refusal to participate in the study and/or lack of signature of a consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with occurrence of an unfavorable outcome between randomization and day 14 | between randomization and day14
  Unfavorable outcome defined by the onset of at least one of the following between randomization and day 14: hospitalization, death or percutaneous O² saturation ≤ 92% in ambient air
Primary outcome of ancillary virological study : evolution of viral load between day 0 and day 14 | between day 0 and day 14
  Ancillary virological study : evolution of viral load between day 0 and day 14, measured by the threshold cycle,Ct, with PCR on naso-pharyngeal swab

SECONDARY OUTCOMES:
The all-cause mortality rate at day 14 | day 14
The all-cause mortality rate at day 28 | day 28
Rate of patients with occurrence of an unfavorable outcome between randomization and day 28 | between randomization and day 28
  Unfavorable outcome defined by the onset of at least one of the following between randomization and day 28: hospitalization, death or percutaneous O² saturation ≤ 92% in ambient air
The rate of use of mechanical ventilation at day 14 | day 14
The rate of use of mechanical ventilation at day 28 | day 28
The Intensive Care Unit admission rate at day 14 | day 14
The Intensive Care Unit admission rate at day 28 | day 28
Number of days of hospitalization for any cause between day 0 and day 14 | between randomization and day 14
Number of days of hospitalization for any cause between day 0 and day 28 | between randomization and day 28
The time to resolution of all COVID symptoms at day 14 | day 14
  Time to resolution of all COVID-19 symptoms : no COVID symptom for at least 48 hours without symptomatic treatment in previous 24 hours
The time to resolution of all COVID symptoms atday 28 | day 28
  Time to resolution of all COVID-19 symptoms : no COVID symptom for at least 48 hours without symptomatic treatment in previous 24 hours
The rate of use of oxygen therapy at day 14 | between randomization and day 14
The rate of use of oxygen therapy at day 28 | between randomization and day 28
The rate of use of secondary antibiotic therapy (after day 2) at day 14 | between randomization and day 14
The rate of use of secondary antibiotic therapy (after day 2) at day 28 | between randomization and day 28
Clinical status at day 14 | day 14
  Clinical status on a 7-point ordinal scale :
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death.
Clinical status at day 28 | day 28
  Clinical status on a 7-point ordinal scale :
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death.
number of serious adverse events at day 14 | day 14
number serious adverse events at day 28 | day 28
number of adverse events at day 14 | day 14
number of adverse events at day 28 | day 28
The rate of patients with treatment withdrawal | day 14
Ancillary virological study : rate of patients with negative viral load at day 8 | day 8
  Ancillary virological study : rate of patients with negative viral load at PCR on naso pharyngeal swab at day 8
Ancillary virological study : rate of patients with negative viral load at day 14 | day 14
  Ancillary virological study : rate of patients with negative viral load at PCR on naso pharyngeal swab at day 14

CONTACTS AND LOCATIONS:
Overall Officials: Julie CHASTANG, Dr, Principal Investigator — Department of General Medicine

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodological sound proposal.